CLINICAL TRIAL: NCT03605004
Title: Adult Patients With Undiagnosed Conditions and Their Responses to Clinically Uncertain Results From Exome Sequencing
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918124; 18-HG-N124
Record Dates: First submitted 2018-07-27; First posted 2018-07-30 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Undiagnosed Disease
Keywords: Genetic Testing; Variant of Uncertain Significance; Uncertainty; Qualitative
MeSH Terms: conditions — Undiagnosed Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Negative: Adult patients with undiagnosed conditions who have received an uninformative negative result from exome sequence.
- VUS: Adult patients with undiagnosed conditions who have received one or more variants ofuncertain significance from exome sequence.

SUMMARY:
Background:

People with conditions that are unknown or hard to diagnose may be helped by a genetic technique. It is called exome sequencing. It helps diagnose disease by unlocking all the data in a person s genetic code. But the results from it are often unclear. Uncertain results can pose problems for doctors and patients. Researchers want to learn more about how people respond when they get uncertain results.

Objective:

To study the psychological and behavioral effects of getting uncertain results from exome sequencing.

Eligibility:

Adults who have:

Had a diagnostic odyssey for at least 6 months. An example is having clinical symptoms but no diagnosis.

And had exome sequencing to try to reach a diagnosis.

Design:

Participants will choose a date and time for their interview. They will sign a form to give consent and authorization.

Participants will fill out 2 forms. One is the Intolerance of Uncertainty Short Form Scale. The other is the Perceptions of Uncertainties in Genome Sequencing Scale.

Both scales ask about what it is like to get clinically uncertain results from exome sequencing. They focus on coping and other behavioral responses.

Participants will have a phone interview. It will last for 45-60 minutes. It will be recorded and transcribed.

At the start of the call, the researcher will review the consent form with the participant. Participants will give data such as race, education, income, and how long they have been looking for a diagnosis.

Participants will read their responses to the 2 scales during the interview.

DETAILED DESCRIPTION:
Patients pursuing exome sequencing in their quest for diagnosis will most often receive a clinically uncertain result. A clinically uncertain result is a result that has some level of objective uncertainty frequently viewed by clinicians in regard to a patient s diagnosis. A clinically uncertain result can be a result that is negative, with no reportable variants, or that includes one or more variants deemed uncertain with regard to the cause of a patient s illness. Clinically uncertain results present challenges to both providers and patients in the forms of disclosing and processing uncertain health information. This exploratory study aims to seek insight into the psychological and behavioral impact of receiving clinically uncertain results from exome sequencing. Semi-structured phone interviews will be conducted with approximately 30-40 adult patients with undiagnosed conditions who have received clinically uncertain result from exome sequencing. The interviews will focus on the experience of receiving the clinically uncertain result, with emphasis on appraisal of uncertainty, coping, and other affective and behavioral responses. Interviews will be transcribed and subjected to thematic analysis. Understanding how patients with undiagnosed conditions respond to clinically uncertain results from exome sequencing may inform providers practices around informed consent for exome sequencing and the disclosure of clinically uncertain results through a greater consideration of patient concerns and challenges with adaptation. This study may also identify implications for interventions to reduce negative effects of receiving uncertain genomic information.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Had endured a diagnostic odyssey of at least 6 months before receiving exome sequencing. A diagnostic odyssey may be defined as:

  * Having a set of clinical symptoms but no diagnosis OR
  * Having a clinical diagnosis of a broad category of disease (i.e. ataxia, muscular dystrophy) but no specific diagnosis OR
  * Having a clinical diagnosis composed of psychosomatic and/or descriptive diagnoses that individually define single symptoms or groups of symptoms (i.e. migraines, IBS, joint pain), but that do not explain the entire phenotype
* and Had exome sequencing in an attempt to attain diagnosis
* and Received post-test counseling for exome sequencing by a genetic counselor
* and Received a clinically uncertain result from exome sequencing. For the purposes of this study, a clinically uncertain result is defined as one of the following options:

  * One or more VUSs
  * A negative test result (no reported variants)
* and Result disclosure for exome sequencing occurred anywhere from 1 week to 7 years prior to being interviewed

EXCLUSION CRITERIA:

* Exome sequencing results provided a genetic diagnosis for the patient that does not fall into one of the above inclusion categories
* Patient was under age 18 at time of clinically uncertain result disclosure
* Patient has a cognitive disability that prevents him/her from comprehensibly answering interview questions
* Patient cannot speak or understand English

Patients who have since received a genetic diagnosis (from some other mechanism besides their exome sequencing test) may still participate in the study if they are able to recount their experiences around receiving this sort of exome sequencing result during the time they were undiagnosed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be received from up to 250 potential participants, in order to do interviews with a sample of approximately 30-40 participants. Participants are adult patients with undiagnosed conditions who have received one of the most common types of clinically uncertain results (negative result or one or more variants of uncertain significance (VUSs) without a known pathogenic result) from exome sequencing. Patients will be recruited from Johns Hopkins Hospital Genetics Clinics and Kennedy Krieger Institute.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Recall and Perception | Interview
  Extent of the patients recall of their clinically uncertain result, including their understanding of the limitations of a clinically uncertain result due to its uncertain nature. It will also explore how patients appraise the uncertainty related to their clinically uncertain result, as well as their perceptions of the relationship between their clinically uncertain result and the cause of their illness.
Affective and Behavioral Responses | Interview
  How patients describe and categorize their emotional reactions to receiving clinically uncertain result from exome sequencing. It will also explore how patients describe their behavior in response to clinically uncertain result disclosures, such as use of coping strategies and decisions to disclose their results to family and friends.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erby, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - Johns Hopkins School of Public Health, Baltimore, Maryland
  - Kennedy Krieger Institute, Baltimore, Maryland

REFERENCES:
- [Background] Vos J, Otten W, van Asperen C, Jansen A, Menko F, Tibben A. The counsellees' view of an unclassified variant in BRCA1/2: recall, interpretation, and impact on life. Psychooncology. 2008 Aug;17(8):822-30. doi: 10.1002/pon.1311. PMID 18157792
- [Background] Han PKJ, Umstead KL, Bernhardt BA, Green RC, Joffe S, Koenig B, Krantz I, Waterston LB, Biesecker LG, Biesecker BB. A taxonomy of medical uncertainties in clinical genome sequencing. Genet Med. 2017 Aug;19(8):918-925. doi: 10.1038/gim.2016.212. Epub 2017 Jan 19. PMID 28102863
- [Background] Skinner D, Raspberry KA, King M. The nuanced negative: Meanings of a negative diagnostic result in clinical exome sequencing. Sociol Health Illn. 2016 Nov;38(8):1303-1317. doi: 10.1111/1467-9566.12460. Epub 2016 Aug 19. PMID 27538589